CLINICAL TRIAL: NCT01769391
Title: A Randomized, Multicenter, Open-Label, Phase 2 Study of Paclitaxel-Carboplatin Chemotherapy Plus Necitumumab (IMC-11F8) Versus Paclitaxel-Carboplatin Chemotherapy Alone in the First-Line Treatment of Patients With Stage IV Squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Necitumumab and Chemotherapy in Participants With Stage IV Squamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14790; I4X-MC-JFCL (Other: Eli Lilly and Company); 2012-003214-13 (EudraCT Number)
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2016-05-05 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Squamous Non Small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: interventions — necitumumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Necitumumab +Paclitaxel+Carboplatin (Experimental): Necitumumab 800 milligram (mg) administered intravenously (IV) on Days 1 and 8 of every 3 week cycle.
  Paclitaxel 200 milligram per square meter (mg/m²) administered IV on Day 1 of every 3 week cycle.
  Carboplatin Area Under the Curve (AUC)6 (mg•min/mL) administered IV on Day 1 of every 3 week cycle.
  The combination of paclitaxel-carboplatin and necitumumab may continue for a maximum of 6 cycles. Necitumumab may continue until Progressive Disease (PD), toxicity requiring cessation, protocol noncompliance, or withdrawal of consent.
  Interventions: Drug: Necitumumab; Drug: Paclitaxel; Drug: Carboplatin
- Paclitaxel + Carboplatin (Active Comparator): Paclitaxel 200 mg/m² administered IV on Day 1 of every 3 week cycle. Carboplatin AUC=6 administered IV on Day 1 of every 3 week cycle. The combination of paclitaxel-carboplatin may continue for a maximum of 6 cycles. After completion of chemotherapy, participants will be followed until radiographic documentation of PD.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Necitumumab — Administered IV
  Other Names: LY3012211; IMC-11F8
  Arms: Necitumumab +Paclitaxel+Carboplatin
Drug: Paclitaxel — Administered IV
Drug: Carboplatin — Administered IV

SUMMARY:
The main purpose of this study is to evaluate if necitumumab added to standard chemotherapy of paclitaxel and carboplatin is more effective to treat cancer than the standard chemotherapy of paclitaxel and carboplatin alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous NSCLC
* Stage IV disease at time of study entry based on American Joint Committee on Cancer (AJCC) 7th edition
* Measurable disease at time of study entry as defined by Response Evaluation Criteria in Solid Tumors, (RECIST) Version 1.1
* Archived or recent tumor tissue (minimum of 5 unstained tissue slides or a paraffin-embedded tissue block) available for analysis of epidermal growth factor receptor (EGFR) protein expression by immunohistochemistry (IHC) and other biomarker assessments

Exclusion Criteria:

* Nonsquamous NSCLC
* Prior anticancer therapy with monoclonal antibodies, signal transduction inhibitors, or any therapies targeting the EGFR, vascular endothelial growth factor (VEGF), or VEGF receptor
* Previous chemotherapy for NSCLC
* Major surgery or received any investigational therapy in the 4 weeks prior to randomization
* Chest irradiation within 12 weeks prior to randomization (except palliative irradiation of bone lesions, which is allowed)
* Brain metastases that are symptomatic or require ongoing treatment with steroids or anticonvulsants (Participants who have undergone previous radiotherapy for brain metastases, who are now nonsymptomatic and no longer require treatment with steroids or anticonvulsants, are eligible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2013-01; Primary Completion 2015-04 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (51):
- United States (33):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jonesboro, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sacramento, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colorado Springs, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fleming Island, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Port Saint Lucie, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. Petersburg, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Macon, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Savannah, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valdosta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kalamazoo, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lansing, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woodbury, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lincoln, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cherry Hill, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hackensack, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Latham, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eugene, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Worth, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Woodlands, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Großhansdorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Immenhausen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
- Mexico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., León
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Poland (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Głuchołazy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olsztyn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Otwock
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Radom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg, Russia
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulsan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A completer is defined as having a complete radiographic assessment at baseline and at least one complete post-baseline radiographic assessment of CR, PR , SD or PD.
Groups:
- Necitumumab +Paclitaxel+Carboplatin: Necitumumab 800 milligram (mg) administered intravenously (IV) on Days 1 and 8 of every 3 week cycle.
  Paclitaxel 200 mg per square meter (mg/m²) administered IV on Day 1 of every 3 week cycle.
  Carboplatin AUC6 administered IV on Day 1 of every 3 week cycle.
- Paclitaxel + Carboplatin: Paclitaxel 200 mg/m² administered IV on Day 1 of every 3 week cycle. Carboplatin AUC6 administered IV on Day 1 of every 3 week cycle. The combination of paclitaxel-carboplatin may continue for a maximum of 6 cycles.
Period: Overall Study
Arm/Group | Necitumumab +Paclitaxel+Carboplatin | Paclitaxel + Carboplatin
Started | 110 | 57
Received at Least One Dose of Study Drug | 106 | 55
Completed | 93 | 48
Not Completed | 17 | 9
Not completed — Death | 10 | 1
Not completed — Adverse Event | 0 | 3
Not completed — Progressive Disease | 1 | 2
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Investigator Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Necitumumab +Paclitaxel+Carboplatin: Necitumumab 800 milligram (mg) administered intravenously (IV) on Days 1 and 8 of every 3 week cycle.
  Paclitaxel 200 milligram per square meter (mg/m^2) administered IV on Day 1 of every 3 week cycle.
  Carboplatin AUC6 administered IV on Day 1 of every 3 week cycle.
- Total: Total of all reporting groups
Arm/Group | Necitumumab +Paclitaxel+Carboplatin | Paclitaxel + Carboplatin | Total
Number analyzed (Participants) | 110 | 57 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (9.36) | 64.7 (8.27) | 65.3 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 13 | 36
  Male | 87 | 44 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 105 | 53 | 158
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 10 | 6 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 97 | 47 | 144
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 28 | 12 | 40
  United States | 53 | 25 | 78
  Poland | 12 | 7 | 19
  South Korea | 10 | 6 | 16
  Mexico | 3 | 3 | 6
  Germany | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve Best Overall Tumor Response of Complete Response (CR) or Partial Response (PR) (Objective Response Rates [ORR])
Description: The denominator of ORR (Objective Response Rate) includes each participant enrolled who received any amount of study drug (necitumumab, gemcitabine, and/or cisplatin), and who had a complete radiographic assessment at baseline and at least one complete radiographic assessment post-baseline. The numerator includes those participants counted in the denominator with a confirmed best overall tumor response of partial or complete response (Complete Response (CR): disappearance of all non-nodal target lesions, with the short axes of any target lymph nodes reduced to <10 millimeters (mm). Partial Response (PR): at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph nodes), taking as reference the baseline sum diameter.) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Time Frame: Baseline to Disease Progression or Death (Up to 24 Months)
Population: All randomized participants that received at least 1 dose of study drug, who had a complete radiographic assessment at baseline and at least 1 complete radiographic assessment post-baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Necitumumab +Paclitaxel+Carboplatin: Necitumumab 800 milligram (mg) administered intravenously (IV) on Days 1 and 8 of every 3 week cycle.
  Paclitaxel 200 milligram per square meter (mg/m²) administered IV on Day 1 of every 3 week cycle.
  Carboplatin Area Under the Curve (AUC)6 (mg•min/mL) administered IV on Day 1 of every 3 week cycle.
Arm/Group | Necitumumab +Paclitaxel+Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 94 | 50
percentage of participants | 48.9 [38.5 to 59.5] | 40.0 [26.4 to 54.8]

2. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from the date of randomization to the date of death from any cause. For participants not known to have died as of the data cut-off date, OS was censored at the last contact date (last contact for participants in post-discontinuation = last known alive date in mortality status).
Time Frame: Randomization to Date of Death (Up to 24 Months)
Population: All randomized participants; (49 and 19 censored participants in Paclitaxel + Carboplatin + Necitumumab and Paclitaxel + Carboplatin Arms, respectively.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Paclitaxel + Carboplatin: Paclitaxel 200 mg/m² administered IV on Day 1 of every 3 week cycle. Carboplatin AUC=6 administered IV on Day 1 of every 3 week cycle. The combination of paclitaxel-carboplatin may continue for a maximum of 6 cycles.
Arm/Group | Necitumumab +Paclitaxel+Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 110 | 57
months | 13.2 [9.7 to 15.9] | 11.2 [8.2 to 12.7]

3. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Necitumumab
Time Frame: Pre-infusion Cycle 1, Day 1; Cycle 3, Day 1; Cycle 5; Day 1 (within 2 hours prior to beginning of infusion)
Population: All participants who received at least one dose of necitumumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (μg/mL)
Groups:
- Necitumumab +Paclitaxel+Carboplatin: Necitumumab 800 milligram (mg) administered intravenously (IV) on Days 1 and 8 of every 3 week cycle.
  Paclitaxel 200 milligram per square meter (mg/m²) administered IV on Day 1 of every 3 week cycle.
  Carboplatin AUC6 administered IV on Day 1 of every 3 week cycle. The combination of paclitaxel-carboplatin and necitumumab may continue for a maximum of 6 cycles.
Arm/Group | Necitumumab +Paclitaxel+Carboplatin
Number analyzed (Participants) | 92
microgram/milliliter (μg/mL)
  Cycle 1, Day 1 (n=92) | 262.418 (32.84)
  Cycle 3, Day 1 (n=72) | 296.843 (62.97)
  Cycle 5, Day 1 (n=62) | 303.475 (53.75)

4. Secondary Outcome: Percentage of Participants With Anti Necitumumab Antibodies
Time Frame: Baseline to End of Cycle 6
Population: All participants who received any amount of necitumumab and had post baseline antibody data.
Measure: Number; unit: percentage of participants
Groups:
- Necitumumab + Paclitaxel+ Carboplatin: Necitumumab 800 milligram (mg) administered intravenously (IV) on Days 1 and 8 of every 3 week cycle.
  Paclitaxel 200 milligram per square meter (mg/m²) administered IV on Day 1 of every 3 week cycle.
  Carboplatin AUC6 administered IV on Day 1 of every 3 week cycle.
Arm/Group | Necitumumab + Paclitaxel+ Carboplatin
Number analyzed (Participants) | 106
percentage of participants | 2.8

5. Secondary Outcome: Progression-Free Survival
Description: Progression-Free Survival (PFS) is defined as the time from randomization until the first radiographically documented progressive disease (PD) or death from any cause. PD defined by Response Evaluation Criteria in Solid Tumors Criteria (RECIST version 1.1) as at least a 20% increase in the sum of the diameters of target lesions,taking as reference the smallest sum on study (including the baseline sum if that is the smallest). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression. For participants not known to have died as of the data cut-off date and who do not have objective PD, PFS will be censored at the date of the last complete radiographic assessment.
Time Frame: Randomization to Progressive Disease or Death (Up to 24 Months)
Population: All randomized participants; with 15 and 7 censored participants in Paclitaxel +Carboplatin + Necitumumab and Paclitaxel +Carboplatin Arms, respectively.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Necitumumab +Paclitaxel+Carboplatin: Necitumumab 800 milligram (mg) administered intravenously (IV) on Days 1 and 8 of every 3 week cycle.
  Paclitaxel 200 milligram per square meter (mg/m²) administered IV on Day 1 of every 3 week cycle.
  Carboplatin AUC6 administered IV on Day 1 of every 3 week cycle.
- Paclitaxel + Carboplatin: Paclitaxel 200 mg/m² administered IV on Day 1 of every 3 week cycle. Carboplatin AUC6 administered IV on Day 1 of every 3 week cycle.
Arm/Group | Necitumumab +Paclitaxel+Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 110 | 57
months | 5.4 [4.2 to 5.7] | 5.6 [4.3 to 6.8]

6. Secondary Outcome: Percentage of Participants Who Achieve Best Overall Disease Response of Complete Response (CR), Partial Response (PR) or Stable Disease (SD) (Disease Control Rate [DCR])
Description: Defined using the same denominator as defined in ORR. Among participants counted in the denominator, the numerator counts those with a confirmed best tumor response of SD, PR, or CR per RECIST 1.1. (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; PR at least 30% decrease in the sum of diameter of target lesions; CR: disappearance of all target lesions).
Time Frame: Baseline to Progressive Disease and/or Death (Estimated up to 24 Months)
Population: All randomized participants who received at least 1 dose of study drug and who had a complete radiographic assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Necitumumab +Paclitaxel+Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 94 | 50
percentage of participants | 87.2 [78.8 to 93.2] | 84.0 [70.9 to 92.8]

7. Secondary Outcome: Percent Change in Tumor Size (CTS)
Description: CTS is defined as maximum percent change from baseline in the sum of target lesions.
Time Frame: Baseline to Progressive Disease or Death (Up to 24 Months)
Population: All randomized participants who received at least 1 dose of study drug and who had a decrease from baseline in the sum of target lesions.
Measure: Mean (Standard Deviation); unit: percent change in tumor size
Arm/Group | Necitumumab +Paclitaxel+Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 83 | 43
percent change in tumor size | -44.3 (22.8) | -38.65 (24.4)

8. Secondary Outcome: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Necitumumab
Time Frame: Cycle 1, Day 8 ; Cycle 2, Day 1; Cycle 3, Day 1;Cycle 4, Day1;Cycle 5, Day 1; Cycle 6, Day 1 (within 2 hours prior to beginning of infusion)
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Necitumumab +Paclitaxel+Carboplatin
Number analyzed (Participants) | 92
nanogram/milliliter (ng/mL)
  Cycle 1, Day 8 (n-85) | 59.269 (59.06)
  Cycle 2, Day 1 (n=79) | 47.874 (79.89)
  Cycle 3, Day 1 (n=76) | 78.142 (70.99)
  Cycle 4, Day 1 (n=70) | 80.392 (74.42)
  Cycle 5, Day 1 (n=62) | 89.137 (88.94)
  Cycle 6, Day 1 (n=59) | 87.043 (85.02)

ADVERSE EVENTS:
Description: All participants who received at least 1 dose of study drug.
Groups:
- Paclitaxel + Carboplatin: Paclitaxel 200 mg/m²) administered IV on Day 1 of every 3 week cycle. Carboplatin AUC6 administered IV on Day 1 of every 3 week cycle. The combination of paclitaxel-carboplatin may continue for a maximum of 6 cycles.
Arm/Group | Necitumumab +Paclitaxel+Carboplatin | Paclitaxel + Carboplatin
Serious Adverse Events (participants affected / at risk) | 43/106 | 21/55
Other Adverse Events (participants affected / at risk) | 102/106 | 49/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Necitumumab +Paclitaxel+Carboplatin (N=106) | Paclitaxel + Carboplatin (N=55)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7) | 2 (3)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 4 (4)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 5 (10) | 0 (0)
Brain death (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 14 (15) | 4 (4)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (4) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Necitumumab +Paclitaxel+Carboplatin (N=106) | Paclitaxel + Carboplatin (N=55)
Anaemia (Blood and lymphatic system disorders) | 34 (87) | 27 (62)
Leukopenia (Blood and lymphatic system disorders) | 9 (16) | 9 (15)
Neutropenia (Blood and lymphatic system disorders) | 37 (73) | 16 (43)
Thrombocytopenia (Blood and lymphatic system disorders) | 27 (67) | 14 (31)
Vision blurred (Eye disorders) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 8 (11) | 2 (2)
Constipation (Gastrointestinal disorders) | 25 (28) | 15 (23)
Diarrhoea (Gastrointestinal disorders) | 26 (34) | 12 (18)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 3 (3)
Nausea (Gastrointestinal disorders) | 27 (35) | 20 (34)
Stomatitis (Gastrointestinal disorders) | 14 (15) | 3 (3)
Vomiting (Gastrointestinal disorders) | 13 (17) | 8 (11)
Asthenia (General disorders) | 18 (31) | 3 (5)
Fatigue (General disorders) | 33 (52) | 24 (48)
Non-cardiac chest pain (General disorders) | 7 (8) | 1 (1)
Oedema peripheral (General disorders) | 11 (15) | 7 (9)
Pain (General disorders) | 7 (9) | 0 (0)
Pyrexia (General disorders) | 10 (16) | 4 (5)
Conjunctivitis (Infections and infestations) | 7 (9) | 0 (0)
Paronychia (Infections and infestations) | 6 (9) | 0 (0)
Pneumonia (Infections and infestations) | 6 (9) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 7 (9) | 0 (0)
Neutrophil count decreased (Investigations) | 8 (18) | 6 (7)
Weight decreased (Investigations) | 31 (49) | 14 (20)
Decreased appetite (Metabolism and nutrition disorders) | 34 (40) | 15 (20)
Dehydration (Metabolism and nutrition disorders) | 11 (15) | 10 (17)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (9) | 3 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 10 (19) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 14 (28) | 4 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 25 (74) | 7 (12)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (13) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (61) | 13 (29)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 8 (14)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 10 (10) | 4 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (9)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (44) | 12 (21)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (10) | 8 (8)
Dizziness (Nervous system disorders) | 14 (16) | 8 (10)
Dysgeusia (Nervous system disorders) | 8 (10) | 4 (4)
Headache (Nervous system disorders) | 4 (6) | 7 (7)
Neuropathy peripheral (Nervous system disorders) | 13 (21) | 9 (18)
Paraesthesia (Nervous system disorders) | 3 (3) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 31 (54) | 13 (24)
Syncope (Nervous system disorders) | 8 (8) | 1 (1)
Anxiety (Psychiatric disorders) | 6 (6) | 0 (0)
Insomnia (Psychiatric disorders) | 14 (16) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (24) | 10 (10)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (29) | 6 (13)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 28 (30) | 10 (11)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 23 (40) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 13 (13) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 22 (69) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (17) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 12 (16) | 0 (0)
Hypotension (Vascular disorders) | 12 (13) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days